CLINICAL TRIAL: NCT05352841
Title: Determination of Salivary Concentrations of Leptin and Adiponectin, Ability to Reduce Ferric Ions and Total Antioxidant Capacity of Saliva in Patients With Early Childhood Caries
Brief Title: Leptin, Adiponectin, FRAP and Tac in Patients With Early Childhood Caries
Acronym: LESSEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Bojan Petrovic, Professor Bojan Petrovic, University of Novi Sad
Other Study IDs: 02-2021
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Early Childhood Caries
Keywords: Total antioxidant capacity; FRAP; Leptin; Adiponectin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caries free children: Children old 72 months or younger with no caries lesion
  Interventions: Diagnostic Test: Salivary sample analysis
- Children with severe form of early childhood caries: Children with severy form of early childhood caries, S-ECC are those having 3 to 5 years , and have more than four, five and six tooth surfaces affected in the primary front teeth at 3, 4 and 5 years, respectively. Caries in children under 3 years of age involving one or more smooth surfaces and in children under 6 years of age affecting one or more smooth surfaces in the front teeth or total dmfs score equal or higher than 6 would be also classified as S-ECC.
  Interventions: Diagnostic Test: Salivary sample analysis

INTERVENTIONS:
Diagnostic Test: Salivary sample analysis — The status of caries will be recorded based on the WHO recommendation, 1997. The children will then be divided into two groups depending on whether they are diagnosed caries (group I) or without carious lesions (group II).After the examination, unstimulated saliva will be collected for analysis (subject to all conditions in proper sampling and without contamination) in a sterile disposable laboratory container with a wide opening and lid. Patients will be asked to tilt their head slightly and not swallow or move their tongue or lips during the collection period. Instructions will be given to accumulate saliva in the mouth for a maximum of 2 minutes and he or she will be asked to spit the accumulated saliva into the receiving court. About 1 ml of unstimulated saliva will be collected.

SUMMARY:
Caries is characterized by the same etiological factors that lead to other chronic non-communicable diseases that are associated with increased dietary sugar intake, such as cardiovascular disease, diabetes and obesity. Early childhood caries is an unacceptable burden for children, families and society. In order to enable the prevention of early childhood caries, it is necessary to actively act on the part of different participants who can influence different aspects of the etiology of caries. Examining the non-specific defense mechanisms of the organism would help shed light on the connection between early childhood caries and other chronic non-communicable diseases, with which they share the same etiological factors.

It is also considered that a child has S-ECC if he is 3 to 5 years old, has more than four, five and six tooth surfaces affected in the primary front teeth at 3, 4 and 5 years, respectively. S-ECC replaces the previous term known as "caries of care bottles". By definition, caries in children under 3 years of age involving one or more smooth surfaces and in children under 6 years of age affecting one or more smooth surfaces in the front teeth or total dmfs score ‡ 6 would be classified as S-ECC. These proposed terms appear to be gaining international acceptance in the current dental literature.

DETAILED DESCRIPTION:
Early childhood caries (ECC) is the most common chronic non-communicable disease in preschool children, and is defined as the presence of one or more carious (uncavitated or cavited) lesions, the absence of one or more teeth (due to caries) or the presence of fillings. any deciduous tooth in a child 72 months of age or younger. Early childhood caries is a disease that is directly dependent on diet. Early childhood caries research is increasingly focused on establishing a link between general and oral health, as well as a local and systemic response to this disease. Antioxidants present in the human body include compounds that act to reduce oxidative stress and the action of free radicals on the human body. It is thought that saliva, through salivary antioxidants, may be the first line of defense against oxidative stress. Salivary antioxidants are a group of enzymes consisting of salivary peroxidase, salivary uric acid, and several smaller enzymes. The combined activity of these enzymes in reducing oxidative stress is often referred to in the literature as Total Antioxidant Capacity (TAC) of saliva. The connection between early childhood caries, rampant caries and increased total antioxidant capacity of saliva has already been described in the literature. Also, the total antioxidant capacity of saliva has been shown to have a linear relationship with age, while no significant dependence has been shown with sex. TAC and Feric Reduction Power (FRAP) have also been studied in patients with periodontitis. Lower TAC and FRAP values in unstimulated and stimulated saliva were confirmed, however, TAC and FRAP concentrations could not be related to the degree and stage of periodontal disease.

Leptin and adiponectin are considered key biomarkers of metabolic dysregulation and comorbidity in both children and adults. Leptin is a polypeptide hormone of 167 amino acids derived from adipocytes, which has been shown to reduce nutrient intake and increase energy expenditure. Its serum concentration is positively associated with total body fat in adults and children. Leptin is a hormone that regulates food intake and energy distribution. It is a protein secreted primarily by fat cells. The salivary glands produce, store and secrete leptin and its level increases with the flow of saliva. A link between leptin levels and tooth loosening during orthodontic treatment has also been found. On the other hand, patients with advanced periodontal disease had lower levels of this hormone. Its role in other diseases of the oral cavity has not been fully investigated. Adiponectin is an adipocyte-derived hormone that regulates glucose and lipid metabolism, improves fatty acid oxidation and insulin sensitivity, and inhibits glucose production in the liver. In addition, adiponectin has strong anti-inflammatory properties. In addition to its previously mentioned local effects, adiponectin in breast milk is involved in the regulation of energy balance regulation and may play a role in the regulation of growth and development in the neonatal period and childhood. Adiponectin is also locally produced in the oral cavity, salivary glands and its level is significantly correlated with plasma levels and as such salivary adiponectin has been used as an alternative to blood tests to measure adiponectin levels.

ELIGIBILITY:
Inclusion Criteria:

* children younger than 72 months
* pediatrician confirmation of apropriate growth and development/weight pattern
* referral from the specialist in pediatric and preventive dentistry

Exclusion Criteria:

* children older than 72 months
* presence of chronic medical, intellectual disability
* acute local or symptomic condition
* report aboout deviation from apropriate growth and development/ weight pattern

Ages: 6 Months to 72 Months | Sex: All
Age Groups: Child
Study Population: 40 patients younger than 72 months. All patients will be presented in writing with the opportunity to participate in a clinical trial and will be asked for written consent. If the parents give written consent, and the child gives oral consent to participate in the study, the usual dental examination will be conducted. For the purposes of the research, no additional questionnaire will be used, but the medical and dental anamnesis will be taken from patients and parents in the usual way. For the purposes of the research, demographic data, dietary habits, medical history, fluoride therapy and the use of drugs and / or vitamin supplements will be detected in particular from the general medical documentation. Also, data will be taken on whether the children have been examined by a pediatrician in the last 6 months and whether a normal pattern of growth, nutrition and general health has been determined.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Salivary levels of TAC in caries free children and children with s ECC | 1 month
  ABTS: Result expressed asTotal Antioxidative Capacity (TAC), unit μg/ml Trolox equivalents
Salivary levels of FRAP in caries free children and children with s ECC | 1 month
  Result expressed as mM Fe equivalents
Salivary levels of leptin in caries free children and children with s ECC | 1 month
  Result expressed in pg / ml
Salivary levels of adiponectin in caries free children and children with s ECC | 1 month
  Result expressed in μg / ml

SECONDARY OUTCOMES:
Interrelationship between FRAP, TAC, leptin and adiponectin in caries free children and children with s ECC | 1 month
  Statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Novi Sad, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No